CLINICAL TRIAL: NCT00303225
Title: A Double-Blind, Randomized, Placebo-Controlled, Ascending Single-Dose, Phase I Trial of the Anti-Orthopoxvirus Compound SIGA-246 in Healthy Volunteers
Brief Title: SIGA-246 to Treat Smallpox
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Jorge A. Tavel, M.D./National Institute of Allergy and Infectious Diseases, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060114; 06-I-0114
Record Dates: First submitted 2006-03-14; First posted 2006-03-15 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-08-04

CONDITIONS: Vaccinia
Keywords: Biodefense; Smallpox; Monkeypox; Vaccinia; Prophylaxis; Healthy Volunteer; HV
MeSH Terms: conditions — Vaccinia; Smallpox; Mpox, Monkeypox

INTERVENTIONS:
Drug: Vaccine: SIGA-246

SUMMARY:
This study will test an experimental antiviral drug called SIGA-246 for use against the smallpox virus (variola). Although smallpox has been universally eradicated, it could possibly be brought back as a bioweapon. In the event of a smallpox attack, it would be best to have an antiviral medication in addition to the smallpox vaccine. SIGA-246 has shown to have activity against other viruses from the same family (orthopoxvirus) that smallpox belongs to.

Healthy volunteers who are 18-50 years of age and are not pregnant or breastfeeding may be eligible for this study. Candidates are screened with a medical history and physical examination, blood and urine tests, and an electrocardiogram.

Participants are randomly assigned to receive a one-time dose of SIGA-246 (either 500 mg, 1000 mg, or 2000 mg) or a placebo (sugar pill) taken by mouth. They report to the clinic in the morning for the following procedures:

* Insertion of intravenous (IV) line in the forearm.
* Blood and urine tests before taking the study drug.
* Drug administration within 30 minutes of eating a light breakfast.
* Blood sampling from the IV line at 30 minutes and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 5 and 6, 10 and 12 hours after taking SIGA-246 to determine how the drug is absorbed, distributed, broken down and excreted. Samples are also collected by needle stick at 24 and 48 hours for the same tests.
* Electrocardiogram at 2 hours and 24 hours after taking SIGA-246.
* 24-hour urine collection after taking the SIGA-246.
* Complete diary card at home for 7 days after taking the SIGA-246.
* Follow-up visits at about 2 weeks and about 4 weeks after taking SIGA-246.
* Checks for health changes or problems at every visit.

DETAILED DESCRIPTION:
Historically, smallpox has been responsible for hundreds of millions of deaths. In 1980 the World Health Organization declared the global eradication of smallpox which was achieved through a surveillance and vaccination program using live virus vaccine. In spite of its eradication, the deliberate use of smallpox as a bioterrorist agent remains a threat. While there is an effective vaccine, there have been concerns regarding vaccine complications which have prevented universal vaccination in the absence of disease exposure. In addition, in the event of a smallpox outbreak vaccination may be ineffective in immunocompromised individuals and in those who were exposed to the virus more than 3 days prior to vaccination. Antiviral therapy may be able to supplement a vaccine, however, there are limitations of the currently available drug options. SIGA-246 is an oral medication that has been shown to be highly active against variola virus and has demonstrated safety in animal models. The primary objective of this study is to assess the safety and tolerability of SIGA-246 at various doses with a secondary objective of evaluating the pharmacokinetics of the drug. To achieve these objectives, 30 healthy volunteers will be enrolled into one of three dosing groups (500 mg, 1000 mg, or 2000 mg) to receive an oral, single dose of SIGA-246 or placebo. In each of the three ascending dosing groups there will be 8 active drug recipients and 2 placebo recipients. Safety of the study agents will be assessed by history, physical, and laboratory evaluations. Pharmacokinetic endpoints include C(max), T(max), t(1/2), AUC, CI and urinary excretion. Urine will be collected in 3 8-hour intervals and serial blood samples will be obtained after study agent administration.

ELIGIBILITY:
* INCLUSION CRITERIA:

A participant must meet all of the following criteria:

1. 18 to 50 years old, inclusive.
2. Available for clinical follow-up for the duration of the study.
3. Able and willing to give written informed consent.
4. In good general health without clinically significant medical history.
5. Be able to refrain from taking any medications for 48 hours after study agent administration.
6. Have adequate venous access.
7. Physical examination and laboratory results without clinically significant findings within the 28 days prior to receipt of study drug (i.e., satisfactorily completed screening).

   Laboratory criteria within 28 days prior to receipt of study drug:
8. Hemoglobin within institutional normal range.
9. WBC within institutional normal range.
10. Absolute neutrophil count (ANC) within institutional normal range.
11. Total lymphocyte count within institutional normal range.
12. Platelets within institutional normal range.
13. ALT (SGPT) within institutional norm range. If the ALT is not within normal limits, it may be repeated once within the 28 days prior to receipt of the study drug.
14. Serum creatinine within institutional normal range.
15. Normal urinalysis defined as negative glucose, negative or trace protein, and negative or trace blood in the urine.
16. Negative beta-HCG pregnancy test (urine or serum) on day of receipt of study drug for women of childbearing potential.
17. The participant or his or her partner has undergone surgical sterlization, or the participant agrees either to be abstinent (i.e., heterosexually inactive) or to consistently use two of the following non-hormonal methods of contraception within the 21 days prior to receipt of the study drug and throughout the duration of the study:

    * Condoms, male or female, with or without a spermicide;
    * diaphragm or cervical cap with spermicide;
    * intrauterine device.

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply:

1. Woman who is breast-feeding or planning to become pregnant prior to or during the 4 weeks of study participation.
2. Volunteer is on any concomitant medications, including over the counter medications or herbal supplements, for 14 days before the administration of the study agent.

   Volunteer has a history of any clinically significant conditions including:
3. Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or intravenous corticosteroids.
4. Diabetes mellitus (type I or II), with the exception of gestational diabetes.
5. History of thyroidectomy or thyroid disease that required medication within the past 12 months.
6. Serious angioedema episodes within the previous three years or requiring medication in the previous two years.
7. Hypertension requiring medication.
8. Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
9. Malignancy that is active, or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study.
10. Seizure disorder other than: 1) febrile seizures under the age of two, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) a singular seizure not requiring treatment within the last 3 years.

    Volunteer has:
11. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.
12. Inability to swallow study medication.
13. Any clinically significant abnormal electrocardiogram findings as determined by the cardiologist in the context of the volunteer's history.
14. Received experimental drug within 30 days of study entry or will participate in any experimental study during the study period.
15. Active illicit drug or alcohol abuse.
16. Any clinically significant lactose intolerance that according to the clinician would be unacceptable for study participation, e.g. lactose intolerance that requires Lactaid or other OTC medications to prevent or alleviate symptoms.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-03-13; Study Completion 2006-08-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States